CLINICAL TRIAL: NCT05553821
Title: Evaluation of the Effect of Cold Pressure Application in the Prevention of Hematoma and Ecchymosis After Percutan Coronary Intervention
Brief Title: Effect of Cold Pressure in the Prevention of Hematoma and Ecchymosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Gülzade Duygun Pamuk, Principal investigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-80558721-050.99-194216
Record Dates: First submitted 2022-04-14; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Clinical Nursing Research
Keywords: nursing, coronary angiography, cold application, comprssion

STUDY DESIGN:
Intervention Model Description: There are two groups in the study. The control group is the normal pressure applied group, the application group is the cold pressure applied group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual pressure group (Active Comparator): A sand bag weighing 3.5-4 kg is applied to the CAG area of this group of patients.
  Interventions: Other: A sand bag
- Cold pressure group (Experimental): A cold sand bag weighing 3.5-4 kg is applied to the CAG area of this group of patients.
  Interventions: Other: Cold sand bag

INTERVENTIONS:
Other: Cold sand bag — A sand bag weighing 3.5-4 kg is applied to the CAG area of patients.
  Arms: Cold pressure group
Other: A sand bag — A sand bag
  Arms: Manual pressure group

SUMMARY:
Coronary Artery Disease (CAD) is the most common cardiovascular system disease. According to the World Health Organization data, CAD ranks first among the top 10 causes of death. According to the 2014 data of the Turkish Statistical Institute (TUIK), deaths due to circulatory system diseases are in the first place with 40.4%, and 39.6% of this is ischemic heart diseases. The prevalence of CAD in Turkey is 12% in women and 14% in men. The diagnosis of CAD is largely made on non-invasive tests. Coronary angiography (CAG) is recommended for definitive diagnosis and detection of coronary stenosis. CAG is defined as the manual delivery of contrast material through a catheter sent to the coronary arteries under fluoroscopy and recording the resulting image on a CD. With special catheters advanced through a plastic sheath called a sheath placed in the access tract, contrast agents are administered separately to the left main coronary (LDA) and right main coronary arteries (RCA), and images of the coronary arteries are taken in multiple positions.

Complications related to diagnostic and therapeutic CAG are rare, but vary according to the patient's condition, operator's experience, and the type of procedure. The most common vascular complications are bleeding, hematoma, ecchymosis, pseudoaneurysm, retroperitoneal hemorrhage, arteriovenous fistula. Preventing complications before they develop is actually shown as the most successful treatment. For this reason, it is recommended to use a small-diameter catheter during CAG, to enter the main femoral artery carefully, to interrupt anticoagulant treatment before the procedure, to apply manual compression to the area for at least 20 minutes after the procedure, and to use percutaneous closure devices, which is another method. After the procedure, pressure is applied with a sandbag, manual compression, and a pneumatic compression device. In the sandbag method, a 3-4.5 kg sandbag is placed after the bleeding is controlled by manual pressure on the femoral region where the intervention is made. During this period, the patient's movements are restricted and he is asked to lie flat on his back. In the use of the pneumatic compression device, a pneumatic compression device (closepad) with a transparent window and balloon incision is placed to maintain the compression on the femoral artery after a short period of manual compression. However, it is not preferred because of the risk of embolism and high cost.

In addition to pressure applications, local cold application is effective in preventing perivascular complications. Cold application controls bleeding by reducing capillary blood flow and capillary permeability by vasoconstriction of arterioles. In addition, it reduces the flow rate of the blood and increases its viscosity, thereby making it coagulate. It controls bleeding by blood coagulation, reduced capillary permeability and metabolic requirements. This situation reduces the development of ecchymosis and hematoma. Considering this information, cold application can be preferred for the prevention of hematoma and ecchymosis, which are the most common complications after CAG, because it is practical, inexpensive and comfort-enhancing. The number of studies in the literature in which cold application and pressure application are used together is limited. Based on this information, the current study was planned to evaluate the effectiveness of cold pressure application for the prevention of hematoma and ecchymosis in the CAG intervention area. The hypotheses of the research; H0: Cold pressure application has no effect on the prevention of hematoma and ecchymosis in the CAG intervention area.

H1: Cold pressure application has an effect on the prevention of hematoma and ecchymosis in the CAG intervention area.

DETAILED DESCRIPTION:
MATERIALS AND METHODS Purpose and type of research This study was planned as a randomized controlled intervention study to evaluate the effect of local cold pressure application on the prevention of hematoma and ecchymosis in patients undergoing CAG via the femoral artery.

Dependent, independent and control variables of the study:

Dependent variables; The dependent variable of this study is the development of bleeding, hematoma and ecchymosis, pain after CAG.

Independent variables; Application of cold pressure applied to patients. Control variables: Patient's age, gender, type of procedure, blood pressure, thrombocyte, Pt, Ptz, INR values, heparin dose administered during CAG (60. IU/kg) Place and time of research The research will be carried out in Eskişehir City Hospital Cardiology and Coronary Intensive Care 1,2 services between Nowember 01, 2021 and June 01, 2022.

Eskişehir City Hospital Cardiology Service: It started to serve in October 2018. In the 24-bed cardiology service, patients with diagnoses such as heart failure, rhythm disorder, and chest pain are generally hospitalized. The number of physicians is 10. The number of nurses is 11.

Eskişehir City Hospital Coronary ICU 1 Service: It started to serve in October 2019. In the 8-bed Coronary Intensive Care 1 Service, patients with diagnoses such as heart failure, arrhythmia, chest pain are generally hospitalized. The number of physicians is 10. The number of nurses is 10.

Eskişehir City Hospital Coronary ICU and 2 Service: It started to serve in November 2018. In the 10-bed cardiology service, patients with diagnoses such as heart failure, arrhythmia, chest pain are generally hospitalized. The number of physicians is 10. The number of nurses is 15.

The standard CAG procedure treatment and follow-up process applied to all patients in Eskişehir City Hospital Cardiology and Coronary Intensive Care 1,2 services are as follows; Standard monitoring and care;

* It is questioned whether the patient has antiplatelet and anticoagulant use.
* The patient who comes to the Angio laboratory is monitored by the nurse. Vital signs are recorded. At the same time, the patient is connected to a defibrillator and defibrillation is provided in case of fatal rhythm.
* Under local anesthesia, an incision is made in the intervention area by the physician, sheath is advanced to the femoral artery, and the coronary arteries are visualized by means of radiopaque material.
* When occlusion or stenosis in the coronary arteries is seen by the physician, balloon and/or stent operation is performed. During these procedures, clarification is provided by using drugs such as heparin, perliganit, clotinab. Sheat extraction is done at the time prescribed by the physician.
* If the coronary arteries are seen as open, sheath is removed and the patient is brought to the service or intensive care unit.
* After sheat extraction, manual compression is done for a minimum of 15 minutes.
* Rolled gauze with a diameter of 5 cm is placed on the intervention area.
* A sandbag is placed on the patient's intervention area and immobilized. The sandbag is kept in the intervention area for 4 hours.
* The patient, whose CAG procedure is completed, is taken to the bed in the ICU or the ward by the nurse, his vital signs are evaluated, an EKG is taken, and the rhythm is followed.
* The intervention area is checked hourly by the nurse in terms of vascular complications, pulse, temperature, color change.
* The time of sheat extraction and sandbag removal, vascular complications in the intervention area and vital signs are recorded by the nurse.
* The treatment ordered by the doctor is applied. The universe and sample of the research The population of the study is the patients who were followed up after CAG in Eskişehir City Hospital Cardiology Service and Coronary Intensive Care 1,2 Services. The sample is the patients who meet the sample selection criteria within the specified population. Sample selection criteria;
* over 18 years old
* Conscious
* Patients who underwent CAG for the first time and/or did not undergo CAG in the last 1 year (it is stated that the recovery period in the femoral intervention area after CAG is completed in 3 months (54). Based on this information, in the study, patients who had CAG before had at least 1 year from CAG. criteria have been determined),
* Platelet values within normal limits,
* Patients treated with 10,000 units or less of heparin during angiography. Exclusion criteria from the study;
* Patients who do not agree to participate in the study and/or want to exit the study while continuing the research,
* Those who developed vascular complications in the region before sheat extraction,
* Those who routinely use anticoagulant drugs,
* Those receiving antithrombotic drug (clotinab) treatment,
* Those with peripheral vascular disease. In determining the number of samples in the study, the sample number was calculated as 210 units, 105 units in the SBG group and 105 units in the NBG, based on the results of the study conducted by Güleser (2011)(55) Data collection method The patients who meet the sampling criteria within the scope of the study will be informed verbally and in writing by the researcher before the CAG procedure and the "Voluntary Consent Form" prepared by the researcher will be signed (Appendix-1). The Individual Identification Form will be filled in by using face-to-face interview technique for all patients. Within the scope of the study, the randomization of the patients who meet the sample selection criteria will be made by an expert independent of the research, using the random numbers method obtained on the computer into two groups [cold pressure group (SBG) and normal pressure group (NBG)]. The specialist will deliver the registration order and the group numbers of the patients in a sealed envelope to the researcher who performed the application.

Procedure In addition to the standard treatment, follow-up and care applied for CAG in Eskişehir City Hospital Cardiology and Coronary Intensive Care services, the steps to be applied for SBG and NBG patients during the research are as follows; Cold pressure application: The following procedures will be applied to the patients in the cold pressure application group;

* The temperature of the cold sandbag to be applied to SBG patients will be kept at 18-20 °C. For this, a sandbag will be placed in the freezer of the refrigerator in the clinic at least 2 hours in advance.
* The surface temperature measurement of the cold sandbag taken out of the freezer will be checked with the surface mode of the thermometer and processed into the KAG follow-up form. In the preliminary application made by us regarding this process, the temperature of the sandbag remaining in the freezer for 2 hours and then removed is 18.1 °C in the 0th minute; 10. 19.3 °C per minute; It was determined that it was 19.5 °C in the 20th minute.
* Cold pressure will be applied for 20 minutes by placing a cold sandbag on the patient's intervention area (56.57),
* After 20 minutes, a cold ice pack will be removed and a room temperature sand bag will be placed. The sandbag at room temperature will be kept in the intervention area for 3 hours and 40 minutes.

Normal pressure application: The following steps will be applied to the patients in the normal pressure application group;

* The sandbag to be used for NBG patients will be kept at room temperature and the surface temperature measurement of the sandbag will be evaluated with the surface mode of the thermometer. The detected heat will be recorded on the KAG tracking form.
* Pressure will be applied to the intervention area of the patients by placing a sand bag at room temperature for 4 hours.

During the study, the treatment plan determined by the doctor will be applied to both groups of patients as specified, and no changes will be made in the treatment plan. Pressure will be applied to both groups of patients for 4 hours, and cold pressure will be applied only to SBG patients for the first 20 minutes. The CAG intervention area of all groups will be monitored and recorded for 24 hours with the CAG follow-up form. According to the CAG follow-up form, in both groups of patients;

* Vital sign monitoring every 15 minutes for the first hour
* Bleeding, hematoma, ecchymosis, pain in the intervention area will be monitored every hour and every 6 hours for the first 6 hours.

Data collection tools Patient identification form (Appendix-2): In the form developed by the researchers according to the literature, there are 13 questions including sociodemographic and disease characteristics (58).

CAG follow-up form (Appendix-3): In the form developed by the researchers according to the literature, there are 12 questions regarding the CAG procedure and post-CAG follow-up (peripheral pulse follow-up, peripheral temperature and color change follow-up, bleeding, ecchymosis, hematoma and pain) (59) .

Sandbag: A sandbag with a height of 23 cm, a width of 14 cm and a weight of 5 kg will be used.

Surface heat meter: It will be measured with the surface mode of Merk brand thermometer.

Roll bandage: 5 cm diameter roll gauze will be used. Patch: It will be used as 10 cm wide and 35 cm long. Analysis of data The data obtained from the patient identification form and CAG follow-up form will be analyzed and reported by a biostatistician independent of the research. Parametric and non-parametric tests will be used in the analysis.

Research endpoint The study is planned to be completed with a total of 210 patients, with at least 105 in each group. When this planned number is reached, the research will end and will take approximately one year.

Ethical approval of the research: Before starting the research, written permission will be obtained from the Eskişehir Osmangazi University Clinical Research Ethics Committee and from the Eskişehir City Hospital where the research will be conducted. Written informed consent will be obtained from patients who want to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* Conscious
* Patients who underwent CAG for the first time and/or did not undergo CAG in the last 1 year (it is stated that the recovery period in the femoral intervention area after CAG is completed in 3 months (54). Based on this information, in the study, patients who had CAG before had at least 1 year from CAG. criteria have been determined),
* Platelet values within normal limits,
* Patients treated with 10,000 units or less of heparin during angiography.

Exclusion Criteria:

* Patients who do not agree to participate in the study and/or want to exit the study while continuing the research,
* Those who developed vascular complications in the region before sheat extraction,
* Those who routinely use anticoagulant drugs,
* Those receiving antithrombotic drug (clotinab) treatment,
* Those with peripheral vascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Assesment of vascular complications and pain | First hour
  Diameters of hematoma and ecchymosis (mm) and score of Visual Analog Scale

SECONDARY OUTCOMES:
Assesment of vascular complications and pain | Sixth hour
  Diameters of hematoma and ecchymosis (mm) and score of Visual Analog Scale
Assesment of vascular complications and pain | Twenty forth hour
  Diameters of hematoma and ecchymosis (mm) and score of Visual Analog Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Eskişehir/Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided